CLINICAL TRIAL: NCT06432153
Title: Tampa Scale of Kinesiophobia for Heart Taiwan Version Validation
Status: Not yet recruiting | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Da-Yeh University (Other)
Responsible Party: Sponsor
Other Study IDs: N_112_0424
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular disease; Kinesiophobia; Scale reliability and validity
MeSH Terms: conditions — Cardiovascular Diseases; Kinesiophobia | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- participant: The only group of participant. Participants are outpatient clinical patients diagnosed with cardiovascular disease.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Participants who receive routine clinical care, without additional intervention from the study

SUMMARY:
Early assessment of kinesiophobia in cardiovascular disease patients is essential. However, measurement tools are scarce for assessing activity fear in cardiovascular disease patients domestically. Currently, the Tampa Scale of Kinesiophobia for the Heart, developed by Bäck et al. (2012), is the most commonly used scale for measuring kinesiophobia among cardiovascular disease patients. As there is no tool available domestically to measure kinesiophobia in cardiovascular disease patients, this research aims to translate, revise, and establish the Taiwanese version of the Tampa Scale of Kinesiophobia for Heart and subsequently verify its reliability and validity for clinical assessment of kinesiophobia among cardiovascular disease patients.

The methodology involves following the translation model by Jones et al. (2001) to translate the Tampa Scale of Kinesiophobia for Heart from the English version to the Taiwan version. Structured questionnaires, including demographic and disease-related information, the Tampa Scale of Kinesiophobia for Heart Taiwan Version, the International Physical Activity Questionnaire, the Six-Minute Walk Test, the Taiwan version of the World Health Organization Quality of Life Questionnaire-BREF, the Hospital Anxiety and Depression Scale, and the Pain Catastrophizing Scale will be used at the cardiological outpatient clinic and inpatient ward of a medical center in Central Taiwan. Patients meeting the study's inclusion criteria and consent to participate in this study will be interviewed. Tampa Scale of Kinesiophobia for Heart Taiwan Version will be examined for content validity, construct validity, internal consistency, and test-retest reliability.

DETAILED DESCRIPTION:
Cardiovascular disease patients may avoid physical activity or exercise due to concerns that engaging in physical activities might exacerbate their heart condition or lead to injury. Interpretation of potential injury as a threat can induce kinesiophobia (fear of movement), causing patients to avoid physical activities, which could negatively impact both their physiological and psychological well-being. Previous research indicates a high prevalence of kinesiophobia among cardiovascular disease patients, and this fear negatively affects their physical activity performance, unwillingness to engage in cardiac rehabilitation, and worse quality of life. Therefore, early assessment of kinesiophobia in cardiovascular disease patients is essential. However, measurement tools are scarce for assessing activity fear in cardiovascular disease patients domestically. Currently, the Tampa Scale of Kinesiophobia for the Heart, developed by Bäck et al. (2012), is the most commonly used scale for measuring kinesiophobia among cardiovascular disease patients. As there is no tool available domestically to measure kinesiophobia in cardiovascular disease patients, this research aims to translate, revise, and establish the Taiwanese version of the Tampa Scale of Kinesiophobia for Heart and subsequently verify its reliability and validity for clinical assessment of kinesiophobia among cardiovascular disease patients.

The objective of this study is to translate, revise, and establish the Taiwanese version of the Tampa Scale of Kinesiophobia for Heart and conduct reliability and validity verification.

The methodology involves following the translation model by Jones et al. (2001) to translate the Tampa Scale of Kinesiophobia for Heart from the English version to the Taiwan version. A longitudinal study design will verify the validity and reliability of the Taiwan version of the Tampa Scale of Kinesiophobia for Heart. Structured questionnaires, including demographic and disease-related information, the Tampa Scale of Kinesiophobia for Heart Taiwan Version, the International Physical Activity Questionnaire, the Six-Minute Walk Test, the Taiwan version of the World Health Organization Quality of Life Questionnaire-BREF, the Hospital Anxiety and Depression Scale, and the Pain Catastrophizing Scale will be used at the cardiological outpatient clinic and inpatient ward of a medical center in Central Taiwan. Patients meeting the study's inclusion criteria and consent to participate in this study will be interviewed. Tampa Scale of Kinesiophobia for Heart Taiwan Version will be examined for content validity, construct validity, internal consistency, and test-retest reliability. The collected data will be analyzed using SPSS/PC version 22.0, and statistical methods such as frequency, percentage, mean, standard deviation, reliability analysis, Pearson correlation, and exploratory factor analysis will be used.

This study aims to translate, revise, and establish the Taiwanese version of the Tampa Scale of Kinesiophobia for Heart and verify its reliability and validity for clinical assessment of Kinesiophobia among cardiovascular disease patients. It also aims to provide insight for future clinical research to analyze related factors further and develop intervention strategies, ultimately enhancing physical activity performance and quality of life and engaging in cardiac rehabilitation for cardiovascular disease patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed with cardiovascular diseases by a specialist, including coronary artery disease, arrhythmia, valvular heart disease, and heart failure, with stable conditions;
* (2) aged 18 or above;
* (3) clear consciousness and able to communicate in Mandarin or Taiwanese;
* (4) willing and consent to participate after being informed of the study purpose and procedures.

Exclusion Criteria:

* (1) cognitive impairment
* (2) psychiatric disorders
* (3) long-term bedridden patients who rely on others for daily activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical patients diagnosed with cardiovascular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-16 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia for Heart | baseline and at the end of the third month
  This scale, developed by Bäck et al. (2012), assesses fear of movement in patients with coronary artery disease. It comprises four dimensions: exercise avoidance, fear of injury, dysfunctional self-perception, and perceived risk of heart problems, with 17 items. Each item is scored on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree), and items 4, 8, 12, and 16 are reverse scored. The total score ranges from 17 to 68, with higher scores indicating greater fear of movement. A TSK Heart score below 37 indicates a low fear of movement, while a score of 37 or higher indicates a high fear of movement. The scale's intra-class correlation coefficient is 0.83, and its internal consistency (Cronbach's alpha) is 0.78 (Bäck et al., 2012).

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | baseline and at the end of the third month
  This study uses the short form of the Taiwan version of the IPAQ, developed in collaboration with Liu Ying-Mei and the World Health Organization. It consists of 7 items assessing physical activity over the past week across work, household chores, transportation, and leisure activities, including time and frequency of walking, moderate and vigorous activities, and time spent sitting. The total physical activity is calculated by multiplying each activity category by its corresponding Metabolic Equivalent (MET), execution time, and activity days. An IPAQ score below 600 indicates low physical activity, 600-3000 indicates moderate physical activity, and above 3000 indicates high physical activity. The scale's content validity is 0.994, and its intra-class correlation coefficient is 0.704 (Liou et al., 2008).
6-Minute Walk Test | baseline and at the end of the third month
  This test is commonly used in clinical settings to assess an individual's exercise capacity and endurance by measuring the distance walked in six minutes. During the test, participants are asked to walk as far as possible along a 30-meter corridor in six minutes. They can rest if they experience difficulty breathing (ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories, 2002).
Taiwan Brief Version of the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) | baseline and at the end of the third month
  Professor Yao Kai-Ping developed this questionnaire after obtaining authorization; this questionnaire assesses the quality of life across four domains: physical health, psychological well-being, social relationships, and environment, with 28 items. Each item is scored on a 5-point scale. Scores for each domain are calculated by averaging the scores of the items within that domain and multiplying by 4. Items 3, 4, and 26 are reverse-scored by subtracting the original score from 6. Higher scores indicate a better quality of life. The internal consistency is 0.91, and the content validity of the domains ranges from 0.51 to 0.64 (Taiwan WHOQOL Group, 2000; Yao Kai-Ping, 2002).
Hospital Anxiety and Depression Scale (HADS) | baseline and at the end of the third month
  This study uses the Chinese version of the HADS, translated by Chen Mei-Ling, initially developed by Zigmond and Snaith (1983). The scale consists of 14 items scored on a 4-point Likert scale (0 to 3), with separate scores for anxiety and depression. Each subscale has a total score range of 0 to 21, with higher scores indicating greater levels of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Ling Chang, MSc, Principal Investigator — Changhua Christian Hospital

IPD SHARING:
Plan to Share IPD: No
No plans to share related information.

REFERENCES:
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Back M, Jansson B, Cider A, Herlitz J, Lundberg M. Validation of a questionnaire to detect kinesiophobia (fear of movement) in patients with coronary artery disease. J Rehabil Med. 2012 Apr;44(4):363-9. doi: 10.2340/16501977-0942. PMID 22366980
- [Result] Cakal B, Yildirim M, Emren SV. Kinesiophobia, physical performance, and health-related quality of life in patients with coronary artery disease. Postepy Kardiol Interwencyjnej. 2022 Sep;18(3):246-254. doi: 10.5114/aic.2022.122892. Epub 2022 Dec 17. PMID 36751297
- [Result] Keessen P, Kan KJ, Ter Riet G, Visser B, Jorstad H, Latour C, van Duijvenbode I, Scholte Op Reimer W. Impact of kinesiophobia on initiation of cardiac rehabilitation: a prospective cohort path analysis. BMJ Open. 2022 Nov 25;12(11):e066435. doi: 10.1136/bmjopen-2022-066435. PMID 36428018
- [Result] Jones PS, Lee JW, Phillips LR, Zhang XE, Jaceldo KB. An adaptation of Brislin's translation model for cross-cultural research. Nurs Res. 2001 Sep-Oct;50(5):300-4. doi: 10.1097/00006199-200109000-00008. PMID 11570715
- [Result] Liou YM, Jwo CJ, Yao KG, Chiang LC, Huang LH. Selection of appropriate Chinese terms to represent intensity and types of physical activity terms for use in the Taiwan version of IPAQ. J Nurs Res. 2008 Dec;16(4):252-63. doi: 10.1097/01.jnr.0000387313.20386.0a. PMID 19061172
- [Result] Lynn MR. Determination and quantification of content validity. Nurs Res. 1986 Nov-Dec;35(6):382-5. No abstract available. PMID 3640358
- See also: WHOQOL BREF — https://www.semanticscholar.org/paper/Development-and-verification-of-validity-and-of-the-Yao-Chung/260271b00a65ac23b1324e52ef1597c13559f95d